CLINICAL TRIAL: NCT00788983
Title: Pulse Oximeter Responses to Multiple Levels of Stable Hypoxia
Brief Title: Induced Hypoxia Study for Validation of SpO2 Accuracy
Status: Completed | Type: Observational
Sponsor: Nonin Medical, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 112008
Record Dates: First submitted 2008-11-07; First posted 2008-11-11 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2008-12

CONDITIONS: Hypoxia
Keywords: Induced hypoxia; Pulse oximeter; Nonin Medical; Verification of SpO2 accuracy
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Validate Non-Motion SpO2 Accuracy from 70%-100% of various pulse oximeter/ sensor combinations and various OEM pulse oximeter modules and sensor combinations during induced hypoxia (desaturation).

DETAILED DESCRIPTION:
The testing is conducted on 12 healthy, consenting, non-smoking subjects in accordance with the IRB approved Protocol. The subjects shall be distributed across both genders and a range of skin tones as equally as practical.

An arterial line will be placed in the radial artery of each subject's right arm, and sensors will be attached to each subject. The subjects will be placed in a semi-supine position and allowed to breathe through a mouthpiece while the nose is blocked with a nose-clip.

Hypoxia will be induced by on each subject, as levels of oxyhemoglobin saturation (between 70% and 100%) are achieved by breathing mixtures of nitrogen, room air and carbon dioxide. Inspired O2 concentration will be adjusted breath-by-breath using a computed saturation, based on end-tidal PO2 and PCO2, as sampled by a mass spectrometer. Predicted levels of oxyhemoglobin saturations will be attained and held stable. At a minimum of sixty seconds into each plateau, a 0.5cc waste blood draw through the arterial line, followed by the first 1.0cc sample blood draw. After approximately thirty additional seconds, the second 1.0cc sample blood draw will be taken. The samples will immediately be analyzed by a Radiometer OSM-3 multi-wavelength co-oximeter and recorded. The SpO2 data from the oximeters will be collected via a laptop computer. Concurrent with the end of each blood draw, a marker will be generated on the laptop computers to identify the event.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers
* Healthy; no known blood disorders
* Finger sizes within the sensor specifications
* Minimum 18 years of age

Exclusion Criteria:

* Artificial nails or fingernail polish

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy, consenting, non-smoking subjects, 18 years or greater, both genders and a range of skin tones
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2008-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
SpO2 Accuracy Verification Study (Arms)of ≤3 between 70 & 100% | During Analysis

CONTACTS AND LOCATIONS:
Overall Officials: Philip E Bickler, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, Induced Hypoxia Lab, San Francisco, California, United States